CLINICAL TRIAL: NCT03861637
Title: Impact of Full Correction of Post-transplant Anemia on the Cardiovascular System and Quality of Life in Renal Transplant Recipients Receiving Erythropoietin Stimulating Agents: a Prospective Randomized Controlled Trial.
Brief Title: Impact of Full Correction of PTA in Renal Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamid Al-Essa Organ Transplant Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VDR/JC/81
Record Dates: First submitted 2019-02-28; First posted 2019-03-04 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Intervention Model Description: comparison of partially corrected vs. fully corrected PTA in renal transplant recipients
Who Masked: Participant
Masking Description: INVESTIGATOR
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- drug : ESA for p correction of PTA (Active Comparator): ESA (Aranesp or mir-CERA) injection 1 mg per kg sc every week for 1 year to correct PTA to level between 12-13g/dl.
  Interventions: Other: ESA for correction of PTA to 12-13g/dl
- ara or cera (Active Comparator): ESA (Aranesp) 1mg/ kg (or equivalent doses) of MIR-CERA injection for 1 year to correct PTA to level between 13-15g/dl.
  Interventions: Other: ESA for correction of PTA to 12-13g/dl

INTERVENTIONS:
Other: ESA for correction of PTA to 12-13g/dl — To assess the impact of full correction of chronic PTA(to near normal values) on cardiovascular system and quality of life in renal transplant recipients with stable graft function using erythropoietin stimulating agents in comparison to partially treated PTA with HB level between 12-13g/dl.
  Other Names: ESA for correction of PTA to 13-15g/dl

SUMMARY:
Background:

Post-transplant anemia (PTA) might be associated cardiovascular morbidity and even increased mortality. Objectives:

We aimed to assess the impact of full correction of chronic PTA on cardiovascular system and quality of life in renal transplant recipients with stable graft function using erythropoietin stimulating agents.

Patient and methods: We enrolled 247 kidney recipients with stable graft function to be assessed for anemia. Eligible patients were randomized to achieve target hemoglobin between 11 to 12 g/dl (group 1, n=183), or 13 to 15 g/dl (in group 2, n=64) using ESA. Monthly clinical and laboratory evaluation of kidney graft function was carried out. Moreover, quality of life (QOL) and echocardiography were assessed at the start and at 12 months.

DETAILED DESCRIPTION:
Two hundred and eighty anemic renal transplant recipients with stable graft function- who are followed up in Hamed Al-Essa organ transplant centre - will be assessed for the possible causes of their anemia. Anemia will be defined as Revised European Best Practice guidelines for anemia in renal tx, a Hb level of <11 g/dl should trigger treatment with ESA.

Drugs:

After patients' assessment for possible causes of anemia, each patient will be managed according to the specific cause of anemia i.e. iron, folic, and vitamin b12 deficiencies will be corrected. If anemia will be improved, we will consider such group of patients as corrected group, but if we failed to find specific cause of anemia we will consider them for ESA. Iron supplementation is permitted in order to maintain serum ferritin in the range 100-800 ng/ml or transferring saturation (TSAT) in the range 20-50%. Medications known to affect Hb concentration-e.g. angiotensin converting enzyme inhibitors (ACEI) & angiotensin receptor blockers (ARBS) - will be maintained at a stable dose if already prescribed at the start of the study.

Patients who fulfilled the following criteria will be included in the study:

Adult renal transplant patients (≥18 years). Informed consent. Stable maintenance subcutaneous darbepoetin alfa therapy with constant dose interval during the last 2 months.

Haemoglobin (Hb) ≥10mg/dL (Hct 32%). Transferrin saturation (TSAT) ≥20% (during the screening phase) Serum ferritin ≥100 ng/mL

We will exclude patients with the following criteria:

Acute or chronic bleeding, or erythrocyte transfusion, within the preceding 8 weeks.

Change in Hb level ≥ 2 g/dL during screening phase. Hemolytic anemia. Recent infection or rejection Diastolic blood pressure >100mmHg or discontinuation of ESA due to hypertension in the 6 months prior to study.

Vitamin B12 or folic acid deficiency. Uncontrolled or secondary hyperparathyroidism. Acute or chronic systemic inflammatory disease and/or C-reactive protein (CRP) >30 mg/L.

Hemodialysis due to the failure of a kidney transplant. Malignancy. Eligible patients will be randomized to either target hemoglobin between 11 to 12 gram/dl (group 1), or target hemoglobin between 13 to 15 gram/dl (group 2). The target HB will be achieved using either darbepoetin α once weekly or once every 2 weeks or equivalent dosage of monthly CERA and the dosage will be adjusted during the titration and evaluation phase according to table 1.

The maintenance dosage of each agent will be modified according to the response (hemoglobin changes). In case of any emergencies, the patient will be managed in Hamed Al-Issa organ transplant Centre 24 hours per day. Mobile of the 1st on-call doctor is ( ); Tel of OTC, ward 1(24826490 &24840300 ext. 4100)".

Randomization:

Patients will be classified according to the maintenance dose of ESA, then they will be sub-grouped into males and females. All patients in each subgroup will be arranged alphabetical using Excel program, and a number will be given to each patient. Patients with odd numbers will serve as group1 while those with even numbers will serve as group 2. Patients' files will be marked with sticker according to the corresponding group to facilitate collection of data.

Methods:

Each patient will be evaluated:

Clinically by history taking and thorough medical examination every month in the outpatient clinic.

By Laboratory investigations which will include:

CBC*, HB electrophoresis, Iron-Ferritin- Transferrin saturation, PT(INR) B12, folic acid levels PTH, CR protein, ESR

* Serum cr., Cr cl, LFT, ca/ph, FBS
* Urinary protein (gm / 24h )
* Drug levels Virology profile (CMV, EBV, Parvovirus ) The radiological investigation using abdominal US, echocardiography and carotid Doppler ultrasound.

Quality of life will be assessed in each patient using 25 and 36 questionnaires at the start of enrollment and by the end of 12 months of achieving the target hemoglobin.

NB.1- * indicates that these test will be every month, while other tests will be only at the initial assessment.

2-Blood samples will be sent to the corresponding laboratory without storage and results will be collected according to the laboratory schedule.

3-As the drugs utilized in such study is available for all patients (Kuwaiti and non-Kuwaiti), we will proceed smoothly. However, some of the laboratory tests will need patients own financial support (especially the non-Kuwaiti).

Data analysis:

Descriptive parameters (mean, standard deviation, median, range, and the number of observations) will be presented for continuous observations.

Frequencies (absolute and percentage) are to be shown for qualitative variables (e.g., sex, ethnicity, Hb values within target ranges and occurrence of adverse events).

The safety population will compromise all patients who received at least one dose of study medication. All patients in the safety population who provided at least one Hb value during C.E.R.A. therapy will be included in the intention-to-treat (ITT) population

ELIGIBILITY:
Inclusion Criteria:

* Patients who fulfilled the following criteria were included in the study:
* Adult renal transplant patients (≥21years),
* Informed consent,
* Stable maintenance subcutaneous ESA therapy with constant dose interval during the last 2 months,
* Haemoglobin (Hb) ≥10mg/dL (Hct 32%),
* Transferrin saturation (TSAT) ≥20% (during the screening phase),
* and serum ferritin ≥100 ng/mL

Exclusion Criteria:

We excluded patients with the following criteria:

* Acute or chronic bleeding, or erythrocyte transfusion, within the preceding 8 weeks. change in Hb level ≥ 2 g/dL during screening phase,
* Hemolytic anemia,
* Recent infection or rejection,
* Diastolic blood pressure >100mmHg or discontinuation of ESA due to hypertension in the 6 months prior to study,
* Vitamin B12 or folic acid deficiency,
* Uncontrolled or secondary hyperparathyroidism,
* Acute or chronic systemic inflammatory disease and/or C-reactive protein (CRP) >30 mg/L,
* Hemodialysis due to failure of a kidney transplant,
* and malignancy

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2015-01-20 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
1 year mortality | 12 months
  number of deaths during 1st year of the study related to full correction of PTA

IPD SHARING:
Plan to Share IPD: Undecided